CLINICAL TRIAL: NCT04321785
Title: Caffeine-induced Effects on Sleep, Cognitive Performance, and Underlying Cerebral Correlates During Adolescence - a Randomised, Placebo-controlled, Double-blind Clinical Study
Brief Title: Effects of Caffeine on Sleep-wake Regulation in Teenagers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carolin Reichert (Other)
Collaborators: Swiss National Science Foundation (Other); Pontificia Universidad Catolica de Chile (Other); University of Liege (Other)
Responsible Party: Sponsor-Investigator, Carolin Reichert, Principal Investigator, Psychiatric Hospital of the University of Basel
Organization: Psychiatric Hospital of the University of Basel (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2017-02118
Record Dates: First submitted 2020-03-17; First posted 2020-03-25 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Adolescence; Caffeine
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Caffeine (Experimental)
  Interventions: Other: Caffeine

INTERVENTIONS:
Other: Placebo — placebo capsule (mannitol)
  Arms: Placebo
Other: Caffeine — caffeine capsule (80 mg of caffeine plus mannitol)
  Arms: Caffeine

SUMMARY:
The aim is to quantify the effects of one dose of caffeine (compared to placebo) on sleep and wakefulness in adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported habitual caffeine consumption: min. 80 mg per month until max 300 mg per week as estimated from mean caffeine content per serving of caffeine containing beverages and food
* Body-Mass-Index: 16.2-25.4
* Informed Consent as documented by signature of participant
* Informed Consent as documented by signature of legal representative

Exclusion Criteria:

* Previous enrollment into the current study
* Investigators' family members, employees or other dependent persons
* Left-handedness
* No normal current health as based on questionnaires, screenings of urine, and examination by the physician in charge
* Drug use: Volunteers must be drug-free for the entire duration of the study, with no history of drug or alcohol dependency.
* Participation in other clinical trials <3 months prior to study begin
* Shift work <3 months prior to study begin
* Transmeridian travel (>2 time zones) <1 month prior to study begin
* Extreme Chronotype (Munich Chronotype Questionnaire [17], MCTQ <2 or >7)
* Short or long sleep duration: subjective sleep duration during schooldays not between 6-10 h (based on MCTQ)
* Inability to follow procedures
* Insufficient knowledge of project language (German)
* Circumstances endangering MRI safety
* Non-compliance with sleep/wake times during ambulatory part (deviation of more than ±1.5 hour from scheduled times)

Ages: 14 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Change of sleep after caffeine intake (vs. placebo) | Nighttime sleep recordings start around 4 hours after caffeine/placebo intake
  Structure and intensity of sleep is measured by polysomnography. We focus on changes in deep sleep.
Change of brain blood-oxygen-level-dependent activity after caffeine intake (vs. placebo) | Start of measurements around 45 minutes once after placebo, once after caffeine
  Using magnetic resonance imaging (MRI), we measure blood-oxygen-level-dependent activity in the brain during a working memory task. How higher blood-oxygen-level-dependent activity can be interpreted depends on behavioral performance.

SECONDARY OUTCOMES:
Change in hormonal profile after caffeine intake (vs. placebo) | Per condition (caffeine and placebo) 8 saliva samples (taken around 250 minutes, 230 minutes, 165 minutes, 115 minutes, 65 minutes and 15 minutes before bedtime, and 490 minutes and 520 minutes after bedtime)
  Hormonal levels are measured in saliva samples. We focus on time of melatonin onset (higher values indicate later time).
Change in subjective sleepiness after caffeine intake (vs. placebo) | Per condition (caffeine and placebo) 8 times (around 250 minutes, 230 minutes, 165 minutes, 115 minutes, 65 minutes and 15 minutes before bedtime, and 490 minutes and 520 minutes after bedtime)
  Sleepiness is measured by a questionnaire (Karolinska Sleepiness Scale, KSS). Higher scores on KSS (range between 1 and 9) represent higher sleepiness.
Change in subjective sleep quality after caffeine intake (vs. placebo) | Per condition around 480 minutes after bedtime
  Subjective sleep quality is measured by the Leeds Sleep Evaluation Questionnaire (LSEQ). Four different scales are evaluated: a) Getting to Sleep (range: 1-100, where lower values represent more difficulties to fall asleep), b) Quality of Sleep (range: 1-100, where lower values represent lower quality), c) Awake Following Sleep (range: 1-100, where lower values represent problems to wake up), and d) Behavior Following Wakening (range: 1-100, where lower values represent more sleepiness after awakening).
Change in working memory performance after caffeine intake (vs. placebo) | Performance is measured 3 times in each condition (around 45 minutes, 180 minutes and 780 minutes after treatment)
  Working performance is measured by accuracy in an n-back task (%of correct responses in 2-back versus 0-back)
Change in viglance performance after caffeine intake (vs. placebo) | Performance is measured 3 times in each condition (around 85 minutes, 200 minutes and 730 minutes after treatment)
  Vigilance performance is measured by reaction time patterns in a psychomotor vigilance task
Change in declarative memory performance after caffeine intake (vs. placebo) | Performance is measured 3 times in each condition (around before 40 minutes before treatment and 210 and 760 minutes after treatment)
  Performance is quantified by assessing the course of the number of words recalled from a list of words (learned before treatment)
Change in pattern separation performance after caffeine intake (vs. placebo) | Performance is measured 3 times in each condition (around 20 minutes before treatment and 220 minutes and 770 minutes)
  Cognitive performance is measured by the lure discrimination index and the recognition performance for repeat items.
Change in mental effort during cognitive performance (working memory) after caffeine intake (vs. placebo) | Mental effort is measured 3 times in each condition (around 70 minutes, 200 minutes and 800 minutes after treatment)
  Mental effort is measured by visual analogue scales targeting satisfaction, concentration, exhaustion and motivation. Scores range from 0-100. Higehr scores indicate higher levels on these scales.
Change in well-being after caffeine intake (vs. placebo) | Per condition (caffeine and placebo) 8 times (around 250 minutes, 230 minutes, 165 minutes, 115 minutes, 65 minutes and 15 minutes before bedtime, and 490 minutes and 520 minutes after bedtime)
  Well-being is quantified as mean of three visual analogue scales targeting tension, mood and physical comfort. Scores range from 0-100. Higher scores indicate better well-being.
Change in cerebral blood flow | once after placebo, once after caffeine (start of measurements around 60 minutes after treatment once after placebo, once after caffeine)
  Using magnetic resonance imaging (MRI), we measure levels of cerebral blood flow in the brain during rest.

OTHER OUTCOMES:
Course of caffeine levels and its metabolites | Per condition (caffeine and placebo) 8 samples (taken around 250 minutes, 230 minutes, 165 minutes, 115 minutes, 65 minutes and 15 minutes before bedtime, and 490 minutes and 520 minutes after bedtime)
  Levels of caffeine and its metabolites are measured in sweat and saliva. Higher values represent higher levels.
Expectancy Questions | After each laboratory part (around 810 minutes after treatment)
  Questions regarding the participant's guess in which condition (caffeine vs placebo) they assume to have taken part (categorical: correct [1] vs incorrect [0]), how sure they are (scores range from 1-10, higher scores indicate higher certainty) and open question on reasons/indications for guess.
Craving for caffeine | Per condition (caffeine and placebo) 8 times (around 250 minutes, 230 minutes, 165 minutes, 115 minutes, 65 minutes and 15 minutes before bedtime, and 490 minutes and 520 minutes after bedtime)
  Craving for caffeine is measured using a visual analogue scale. Scores range from 0-100. Higher scores inidicate higher craving.

CONTACTS AND LOCATIONS:
Overall Officials: Carolin Reichert, Principal Investigator — Centre for Chronobiology, Basel
Locations (1):
- Centre for Chronobiology, Basel, Switzerland